CLINICAL TRIAL: NCT07244185
Title: The Effect of Osseodensification and Conventional Implant Site Preparation on Implant Stability of Tapered and Cylindrical Dental Implants
Brief Title: Comparison of Osseodensification and Conventional Drilling on the Stability of Tapered and Cylindrical Implants.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Worood Adnan Akram (Other)
Collaborators: Teaching Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Worood Adnan Akram, The Effect of Osseodensification Versus Conventional Implant Site Preparation on the Primary Stability of Tapered and Cylindrical Dental Implant, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 974124-2024
Record Dates: First submitted 2025-11-13; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Tooth Absence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tapered implant with conventional preparation (Experimental): The osteotomy will be performed following the manufacturer's standard drilling sequence without osseodensification.
  This group will serve to evaluate the effect of conventional implant site preparation on the primary and secondary stability of tapered implants
  Interventions: Procedure: Dental Implant Placement with Osseodensification or Conventional Drilling
- tapered with osseodensification (Experimental): The osteotomy will be prepared with densifying burs operated in a non-subtractive, counterclockwise direction to compact and preserve bone tissue.
  This approach aims to enhance bone density and improve the primary and secondary stability of the tapered implants
  Interventions: Procedure: Dental Implant Placement with Osseodensification or Conventional Drilling
- cylindrical implant with conventional preparation (Experimental): The osteotomy will be performed following the standard sequential drilling protocol recommended by the manufacturer, without applying osseodensification.
  This group will be used to assess the effect of conventional implant site preparation on the primary and secondary stability of cylindrical implants
  Interventions: Procedure: Dental Implant Placement with Osseodensification or Conventional Drilling
- cylindrical with osseodensification (Experimental): The osteotomy will be performed using densifying burs in a non-subtractive, counterclockwise direction, which compacts and preserves the surrounding bone tissue.
  This method is intended to increase bone density and improve both primary and secondary implant stability for cylindrical implants
  Interventions: Procedure: Dental Implant Placement with Osseodensification or Conventional Drilling

INTERVENTIONS:
Procedure: Dental Implant Placement with Osseodensification or Conventional Drilling — Placement of tapered or cylindrical dental implants using osseodensification (bone-compacting technique) or conventional drilling to evaluate implant stability.

SUMMARY:
The effect of osseodensification versus conventional implant site preparation on implant stability for tapered and cylindrical dental implants.

DETAILED DESCRIPTION:
Dental implant stability is a key factor influencing the success of osseointegration and the long-term prognosis of implant-supported restorations. The stability of an implant can be divided into two phases: primary stability, which depends on the mechanical engagement between the implant and the surrounding bone at the time of placement, and secondary stability, which develops through biological bone remodeling and osseointegration over time.

Traditional (conventional) drilling techniques used for implant site preparation are subtractive in nature, meaning they remove bone to create space for the implant. However, this process may reduce bone density at the osteotomy walls, particularly in low-density bone, potentially compromising initial stability.

Osseodensification (OD) is a relatively new, non-subtractive drilling technique introduced by Huwais and colleagues. Instead of removing bone, OD uses specially designed, counterclockwise rotating burs (Densah burs) that laterally compact and densify bone along the walls of the osteotomy.

mplant macrodesign-particularly whether the implant is tapered or cylindrical-also influences stability outcomes.

Tapered implants typically provide higher primary stability due to their wedging effect and better adaptation in underprepared osteotomies, especially in soft bone.

Cylindrical implants, while providing more uniform stress distribution, may rely more heavily on bone density and precise site preparation for achieving optimal stability.

ELIGIBILITY:
Inclusion Criteria:

* 1-Patients who are willing to comply with the study and give their consent. 2-Ability to tolerate conventional surgical and restorative procedure. 3- Healthy patients over 18 years of either gender, having single or multiple missing teeth in the maxilla and/or mandible

Exclusion Criteria:

1. Active infection or inflammation in implant area or neighboring zone.
2. Systemic conditions (medically compromised patient) such as uncontrolled diabetes, coagulation disorders, immune compromised patient, patient treated with bisphosphate drugs, psychiatric problems or unrealistic expectations, pregnant women, any medical condition that affect bone healing.
3. Clinical evidence of parafunctional habits.
4. Active periodontitis.
5. Heavy smokers (≥20 cigarettes a day).
6. Advanced and complicated cases.
7. Patients who not able to follow the treatment protocol or lost during the study period.
8. Patient with history of radiotherapy to the head and neck -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
primary stability | at the time of surgery
  Primary stability refers to the mechanical stability of a dental implant (or any bone implant) immediately after placement, before bone healing or osseointegration occurs.
  It mainly depends on bone quality and density, implant design, and surgical technique.it measured using the osstell through Resonance Frequency Analysis,Higher ISQ values indicate greater primary stability.more than 70 ISQ is considerd high stability.
  Achieving good primary stability is crucial for implant success, as it helps prevent micromovements and supports proper secondary (biological) stability during healing,

SECONDARY OUTCOMES:
secondary stability | after 12 weeks
  Secondary stability refers to the biological stability of a dental implant that develops over time through osseointegration, the direct structural and functional connection between the implant surface and surrounding bone.
  Unlike primary stability, which is mechanical, secondary stability results from bone healing, remodeling, and new bone formation around the implant ..it measured using the osstell through Resonance Frequency Analysis,Higher ISQ values indicate greater stability.more than 70 ISQ is considerd high stability.

CONTACTS AND LOCATIONS:
Locations (1):
- university of baghdad college of dentistry Teaching hospital, Baghdad, Baghdad Governorate, Iraq